CLINICAL TRIAL: NCT05339464
Title: Ready and Healthy for Kindergarten- Pilot Study
Brief Title: Ready and Healthy for Kindergarten
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manuel E. Jimenez, MD, MS, Assistant Professor of Pediatrics & Family Medicine and Community Health, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2021001575; R18HS028574 (AHRQ)
Record Dates: First submitted 2022-04-08; First posted 2022-04-21 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Parenting; Language Development; Literacy; Health Behavior
Keywords: Early literacy; Language development; Family literacy; Bilingualism; Community engagement
MeSH Terms: conditions — Literacy; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family wellness program- Group 1 (Experimental): This group will begin the family wellness program first; approximately, 5 weeks before group 2. The family wellness program consists of 8 parent-child workshops and text message reminders.
  Interventions: Other: Family Wellness program
- Family wellness program- Group 2 (Experimental): This group will begin the family wellness program approximately 5 weeks after group 1.The family wellness program consists of 8 parent-child workshops and text message reminders.
  Interventions: Other: Family Wellness program

INTERVENTIONS:
Other: Family Wellness program — Weekly one-hour online workshops over an 8 week period. Families will also receive text message reminders as part of the intervention.

SUMMARY:
This study pilot tests a family wellness program that promotes academic and physical readiness for school among Latino dual language learners using a mixed methods and community engaged approach.

DETAILED DESCRIPTION:
The investigators propose a pilot randomized controlled trial with wait list control to pilot test a family wellness program designed for Latino dual language learners entering Kindergarten and their families. The investigators will recruit up to 48 parent-child dyads to participate in the study. Families will be randomly assigned to session one beginning in June 2022 or session two beginning in July 2022. The investigators will examine the feasibility and acceptability of the family wellness program as well as preliminary effects on parenting behaviors and child language and literacy skills.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child entering Kindergarten (4-6 years old),
* Primary caregiver identifies as Hispanic/Latino/Latinx,
* Family speaks Spanish at home,
* Cell phone ownership,
* Willing to receive texts, and
* Willing to accept randomization

Exclusion Criteria:

* Children with multiple congenital anomalies or genetic disorders and previously identified developmental delays will be excluded.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Number of sessions attended | 2months
  Number of sessions attended by participants will be used to assess the feasibility of the online family wellness program.
Acceptability assessed by the Acceptability of Intervention Measure (AIM) | 2 months
  Data on perceived acceptability will be captured via parent report on the AIM survey. The AIM is a 4 item survey that assesses acceptability. Higher scores indicate higher acceptability.

SECONDARY OUTCOMES:
Home learning environment | Enrollment, 2months, 4months
  The home learning environment will be assessed with the StimQ, a caregiver-reported measure of cognitive stimulation for children that includes domains on the home literacy environment (READ scale) and responsiveness (Parental Verbal Responsiveness scale). The READ scale includes 3 subdimensions (Book Reading Quantity, Diversity of Content, Book Reading Quality). Scores on the READ scale range from 0 to 18. The Parental Verbal Responsiveness scale includes a subdimension on responsiveness during routines (Everyday Routines). Scores range from 0 to 8. Higher scores indicate more cognitive stimulation
Child vocabulary | Enrollment, 2months, 4months
  Child vocabulary will be assessed using an investigator developed measure. Higher scores indicate higher skills
Child literacy skills | Enrollment, 2 months, 4 months
  Literacy skills including concepts about books, story retelling, narrative thematic knowledge, letter and sound identification will be assessed using an investigator developed measure. Higher scores indicate higher skills
Home health routines | Enrollment, 2 months, 4 months
  Descriptive survey examining health routines including nutrition, physical activity, and sleep

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Jimenez, MD, MS, Principal Investigator — Rutgers University
Locations (1):
- Child Health Institute, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified quantitative data and associated documentation may be made available to users conducting non-profit research under a written data-sharing agreement
Supporting Information: Study Protocol
Time Frame: Data will become available after the study is completed and primary study findings are published in peer-reviewed journals for 10 years after study completion.
Access Criteria: Researchers from accredited institutions may request access to the data for non-profit research. Permission and access will be granted on an ad hoc basis. Only deidentified data will be made available.